CLINICAL TRIAL: NCT02872038
Title: A Multicenter, Randomized, Controlled Trial Comparing Cefepime Monotherapy Versus Combination of Cefazolin Plus Ceftazidime for Empirical Treatment of CAPD-associated Peritonitis
Brief Title: Comparing Cefepime Versus Cefazolin Plus Ceftazidime for CAPD-associated Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: The Kidney Foundation of Thailand (Unknown); Siam Pharmaceutical Co Ltd (Unknown)
Responsible Party: Principal Investigator, Thidarat Kitrungphaiboon, MD, Fellow of Nephrology, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MONOCEF
Record Dates: First submitted 2016-07-25; First posted 2016-08-18 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Peritoneal Dialysis Associated Peritonitis
MeSH Terms: interventions — Cefepime; Cefazolin; Ceftazidime; Control Groups

ARMS (2):
- Treatment (Experimental): Cefepime intraperitoneal continuous dosing
  Interventions: Drug: Cefepime
- Control (Active Comparator): Cefazolin plus Ceftazidime intraperitoneal continuous dosing
  Interventions: Drug: Cefazolin plus Ceftazidime

INTERVENTIONS:
Drug: Cefepime — Cefepime intraperitoneal continuous dosing
  Arms: Treatment
Drug: Cefazolin plus Ceftazidime
  Other Names: Control group
  Arms: Control

SUMMARY:
The purpose of this study is to compare the efficacy of empirical antibiotics of CAPD-associated peritonitis with intraperitoneal, continuous dosing of cefepime monotherapy versus combination of cefazolin and ceftazidime. Patients were randomized to be administered either intraperitoneal cefepime 1 g loading then 250 mg all exchanges (treatment group) or cefazolin and ceftazidime (control group) in the same dose.

DETAILED DESCRIPTION:
The International Society of Peritoneal Dialysis (ISPD) guideline suggest to use combination of antibiotics to cover both of gram positive and gram negative bacteria. The usual regimen in Thailand is cefazolin plus ceftazidime. Despite combination therapy, monotherapy is also possible for empirical treatment of CAPD-associated peritonitis since it helps to lowering staff burden and lowering risk of contamination. Cefepime could be an ideal antibiotic for empirical treatment of CAPD-associated peritonitis as it is an extended-spectrum cephalosporin, forth generation, covering most of gram positive and gram negative bacteria. In addition, cefepime is not broken down by many of the beta-lactamases and less beta-lactamases inducer. This study aims to prove the noninferiority of cefepime monotherapy to cefazolin plus ceftazidime for empirical treatment of CAPD-associated peritonitis.

CAPD-associated peritonitis was diagnosed by at least two of the following criteria: abdominal pain or cloudy peritoneal dialysis fluid (PDF); PDF white cell count > 100/μL with > 50% polymorphonuclear(PMN); and positive gram stain or culture. The patients were randomized into two groups by block of four randomization, sealed envelope. Treatment group was treated with intraperitoneal (IP) cefepime 1 g loading following by maintenance dose 250 mg IP all exchanges. Control group was treated with cefazolin 1 g IP loading and ceftazidime 1 g IP loading following by maintenance dose of cefazolin and ceftazidime 250 mg IP all exchanges. If a patient had residual urine ≥ 100 ml/day, dose of antibiotics would be increased by 25%.

On the first day, the initial blood tests for complete blood count, electrolyte, BUN, creatinine, calcium, phosphate and magnesium were obtained. While peritoneal dialysis fluid were collected using two methods of bacterial culture, both of centrifugation of 50 ml peritoneal dialysis fluid at 3,000 g for 15 minutes and bedside 5-10 ml of peritoneal dialysis fluid inoculated into the blood culture bottles. PDF gram stain and bacterial culture were done. The patients were followed on day 3, 5, 10, 14, 21 and 28 days after the completion of antibiotic course. If clinical improved, the antibiotics would be adjusted according to the culture result and sensitivity after day 5. If clinical not improved the antibiotics would be step up and Tenckhoff catheter removal was considered (on any day of treatment). The patients were treated at least 14 days or 21 days depend on the culture result (as the recommendation of ISPD guideline 2010).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* CAPD initiation more than 4 weeks

Exclusion Criteria:

* Exit site or tunnel infection
* Sepsis
* Previous CAPD-associated peritonitis treatment within 4 weeks
* Drug allergy to cephalosporin
* Tenckhoff catheter malfunction
* Hospitalization more than 48 hours
* Fungal or Mycobacterium infection
* Suspected secondary peritonitis
* Concomitant antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Primary response rate | day 10 of treatment
  Resolution of clinical peritonitis and peritoneal dialysis fluid WBC < 100 /μL with PMN < 50% at day 10

SECONDARY OUTCOMES:
Initial response rate | day 5 of treatment
  Resolution of clinical peritonitis and peritoneal dialysis fluid WBC < 100 /μL with PMN < 50% at day 5

OTHER OUTCOMES:
Complete cure rate | 28 days after completion of antibiotics
  Complete resolution without relapse or recurrent within 28 days after completion of antibiotics.
Relapse peritonitis rate | 28 days after completion antibiotics
  Recur of peritonitis with the same organism or sterile culture within 28 days after completion antibiotics
Recurrent peritonitis rate | 28 days after completion antibiotics
  Recur of peritonitis with different organism within 28 days after completion antibiotics
Death rate | 28 days after completion antibiotics
  Death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Kitrungphaiboon T, Puapatanakul P, Chuengsaman P, Tiskajornsiri K, Halue G, Siribamrungwong M, Matayart S, Chongthanakorn K, Poonvivatchaikarn U, Boonyakrai C, Somboonsilp W, Katavetin P, Praditpornsilpa K, Eiam-Ong S, Johnson DW, Kanjanabuch T. Intraperitoneal Cefepime Monotherapy Versus Combination Therapy of Cefazolin Plus Ceftazidime for Empirical Treatment of CAPD-Associated Peritonitis: A Multicenter, Open-Label, Noninferiority, Randomized, Controlled Trial. Am J Kidney Dis. 2019 Nov;74(5):601-609. doi: 10.1053/j.ajkd.2019.05.011. Epub 2019 Jul 19. PMID 31331757